CLINICAL TRIAL: NCT01191567
Title: Negative Pressure Wound Therapy. Therapy Effects and the Impact on the Patient's Quality of Life
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitement speed
Sponsor: Karolinska Institutet (Other)
Collaborators: Stockholm South General Hospital (Other)
Responsible Party: Principal Investigator, Ann-Mari Wallin, RN, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008/2023-31
Record Dates: First submitted 2010-08-26; First posted 2010-08-31 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Wounds
Keywords: acute wounds; postoperative wounds
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional treatment (Active Comparator)
  Interventions: Procedure: Conventional treatment
- VAC treatment (Experimental)
  Interventions: Procedure: VAC treatment

INTERVENTIONS:
Procedure: VAC treatment — wound treatment with VAC-therapy
  Arms: VAC treatment
Procedure: Conventional treatment — wound treatment with conventional treatment according to the hospitals local routines
  Arms: Conventional treatment

SUMMARY:
Wounds have long been a source of suffering for unfortunate victims and in recent years new complementary methods have been developed in areas where traditional wound treatment has been insufficient. Treating wounds with negative pressure, Vacuum assisted closure® [VAC], is a relatively new method of treatment and knowledge about its effect on patients is limited.

Earlier studies haven't been able to answer the question about which groups of patients that are in most favour of the treatment and what impact the treatment has on the patient's quality of life.

It is important with further research since an effective and mild wound treatment can decrease suffering and increase quality of life for the patient. Wound treatment that does not lead to an achieved treatment goal can lead to a risk for the patient and should be avoided.

The project consists of 4 part studies: Study 1 and 2 are chart review studies of a consecutive series of patients treated with VAC at Södersjukhuset during a 3 year period. The patients are described on the basis of medical, surgical and demographical factors. Outcome is treatment results and risk factors for a treatment failure.

Study 3 and 4 are clinical randomised studies with the aim of studying whether treatment with VAC provides a faster and more effective healing of acute and postoperative wounds, and in what way the treatment affect the quality of life and pain of the patients, compared to conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* acute wounds with substance defect after primary suture demanding further treatment or wounds not primary sutured
* wounds with osteosynthesis, bone or tendon visual regardless wound size
* postoperative infections with wound and substance defect demanding further treatment.
* fasciotomy on extremity

Exclusion Criteria:

* wound size < 2 cm and depth < 1 cm
* pressure ulcers, open abdomen and chronic ulcers
* patients with dementia or mental illness so severe that participation in the study is impossible
* patients non in command of the swedish language
* ongoing treatment with warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
treatment results | 2 weeks
  successfully treated or non-successfully treated
wound size | 2 weeks
  meassured with Visitrak
Quality of life | 2 weeks
  meassured with EQ-5D form and a diary with content analysis

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 2 weeks
costs for treatment | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Södersjukhuset, Stockholm, Sweden